CLINICAL TRIAL: NCT00778076
Title: The Biomechanical Impact of Intra-Articular Hyaluronic Acid in Knee Osteoarthritis Patients: A Randomized, Double Blind, Placebo Controlled Study
Brief Title: The Impact of Hyaluronic Acid Injections on Osteoarthritic Knee Mechanics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Dr. Robert Petrella, The University of Western Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB#: 14017
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee OA, Hyaluronic acid, Gait, Pain, Synovial fluid
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HAG (Active Comparator): Patients that will receive a Hyaluronic acid treatment course consisting of 3 consecutive injections one week apart.
  Interventions: Device: Hyaluronic acid
- PG (Placebo Comparator): Those patients that receive 3 consecutive placebo injections one week apart.
  Interventions: Device: Placebo (Saline injection)

INTERVENTIONS:
Device: Hyaluronic acid — 3 consecutive injections, each one week apart, of 20mg/2ml Hyaluronic acid.
  Other Names: Suplasyn; Sodium Hyaluronate
  Arms: HAG
Device: Placebo (Saline injection) — 3 consecutive injections, each one week apart, of 20mg/2ml of Placebo.
  Other Names: Sham injection; Saline injection
  Arms: PG

SUMMARY:
The purpose of this study is to determine the impact of a regular course of treatment with Hyaluronic acid (HA) injections on gait in knee osteoarthritis (OA) patients. Three consecutive HA injections will be compared to three consecutive placebo injections to determine whether HA's analgesic effect is greater than that of a placebo injection, and to observe whether HA's viscoelastic properties are manifested in a human knee OA population. We hypothesize that HA injections will relieve pain to a greater extent than placebo injections in knee OA patients, and will afford them with improved walking characteristics, such as increased walking speed, and step length.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a severely debilitating disease associated with stiffness and pain in the knee joint, and with a loss of function. Hyaluronic acid (HA) injections are incorporated into non-surgical standard of care for knee OA patients and have been proven to relieve pain in patients who have not received symptomatic relief with other knee OA interventions. HA allows synovial fluid to act as a lubricant and shock absorber for joints, and although this is encouraging ground to advocate for the use of HA treatment in knee OA patients, these properties have yet to be proven in a controlled clinical trial setting. Therefore, we are undertaking this study to observe whether the physiological adaptation in the OA knee joint, initiated by HA injection, will result in biomechanical improvements in human knee OA patients, specifically walking mechanics.

ELIGIBILITY:
Inclusion Criteria:

* 60 - 80 years old.
* Mild to moderate knee osteoarthritis:
* Clinical diagnosis (symptoms).
* Radiographic diagnosis (Kellgren-Lawrence grade I - III).
* Must provide provide informed consent and knowledge of all possible benefits and possible adverse events.
* Available for duration of the study.
* Not taking any other knee osteoarthritis medications during the study.

Exclusion Criteria:

* Non - OA arthritides.
* Hip, ankle, or foot OA.
* End stage OA.
* Lower back/extremity pathology.
* Previous surgery on knee affected by OA (except arthroscopy within the past 12 - 18 months).
* Neurological/Cardiovascular gait impairment.
* Pregnant.
* Cognitively impaired.
* Not available for duration of study.
* Taking other knee OA medications at time of study.
* Gastro-intestinal disturbance.
* Avian allergy or any other contraindication to intra-articular injections with Hyaluronic acid.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Gait analysis with GAITRite software. | Baseline; after each injection; 3 and 6 months post treatment.

SECONDARY OUTCOMES:
WOMAC OA index (pain, stiffness, function); Six minute walk test (function). | Baseline; after each injection; 3 and 6 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Petrella, MD, PhD, Principal Investigator — The University of Western Ontario; Joseph E DeCaria, BA, MSc('09), Study Director — The University of Western Ontario
Locations (1):
- St. Joseph's Health Care, Parkwood Hospital, Aging Rehabilitation and Geriatric Care research center, London, Ontario, Canada

REFERENCES:
- [Background] Tang SF, Chen CP, Chen MJ, Pei YC, Lau YC, Leong CP. Changes in sagittal ground reaction forces after intra-articular hyaluronate injections for knee osteoarthritis. Arch Phys Med Rehabil. 2004 Jun;85(6):951-5. doi: 10.1016/j.apmr.2003.08.095. PMID 15179649
- [Derived] DeCaria JE, Montero-Odasso M, Wolfe D, Chesworth BM, Petrella RJ. The effect of intra-articular hyaluronic acid treatment on gait velocity in older knee osteoarthritis patients: a randomized, controlled study. Arch Gerontol Geriatr. 2012 Sep-Oct;55(2):310-5. doi: 10.1016/j.archger.2011.11.007. Epub 2011 Dec 9. PMID 22169699